CLINICAL TRIAL: NCT00019539
Title: Phase II Randomized Study of Monoclonal Antibody VEGF in Patients With Unresectable Advanced Renal Cell Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066669; NCI-98-C-0159; NCI-T98-0035; NCT00001707 (obsolete NCT alias)
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Stage IV Renal Cell Cancer; Recurrent Renal Cell Cancer
Keywords: adult solid tumor; body system/site cancer; cancer; kidney tumor; kidney/urinary cancer; recurrent renal cell cancer; renal cell cancer; solid tumor; stage IV renal cell cancer; stage, renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Urologic Neoplasms | interventions — Bevacizumab; Thalidomide

INTERVENTIONS:
Drug: bevacizumab
Drug: thalidomide

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them.

PURPOSE: Randomized phase II trial to determine the effectiveness of monoclonal antibody therapy in treating patients who have advanced kidney cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of monoclonal antibody VEGF on time to progression, angiogenesis, and overall survival in patients with unresectable advanced renal cell cancer.

II. Evaluate serum antibody levels and biologically active vascular endothelial growth factor levels in the plasma of patients treated with this regimen.

III. Evaluate the toxicity of this regimen in these patients.

PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by prior interleukin-2 therapy (yes vs no).

Patients are randomized to receive either placebo or one of two doses of monoclonal antibody VEGF. Following an initial loading dose, patients receive one dose of the study drug intravenously every 2 weeks for up to 2 years in the absence of disease progression. Patients who are given placebo and experience disease progression are offered monoclonal antibody VEGF and thalidomide if there are no contraindications.

PROJECTED ACCRUAL:

A total of 150 patients will be accrued for this study over 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically proven unresectable advanced renal cell cancer Measurable disease Must have received or not be a suitable candidate for interleukin-2 therapy No papillary or collecting duct renal cell cancer No CNS metastases --Prior/Concurrent Therapy-- Biologic therapy: See Disease Characteristics No prior thalidomide At least 4 weeks since other prior biologic therapy No other concurrent biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior endocrine therapy No concurrent corticosteroid therapy Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics --Patient Characteristics-- Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 6 months Hematopoietic: WBC at least 1,000/mm3 Platelet count at least 75,000/mm3 No coagulation disorder, active bleeding, or wound healing problem Hepatic: Total bilirubin no greater than 2.0 mg/dL (for patients with Gilbert's disease, direct bilirubin less than 0.5 mg/dL) SGOT or SGPT no greater than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No coronary artery disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No clinically evident preexisting peripheral neuropathy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Chung-Yin Yang, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States